CLINICAL TRIAL: NCT03892733
Title: Improving the Impact of Calorie Labeling Policies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011-579
Record Dates: First submitted 2019-03-15; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Obesity; Diet Habit
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): CHEKS (calorie health, education, knowledge and skills) intervention will educate participants about calories in fast-food and teach skills to select lower calorie fast-food items.
  Interventions: Behavioral: calorie health education knowledge and skills
- Control (No Intervention): Participants will receive a brochure about healthier choices in fast-food restaurants.

INTERVENTIONS:
Behavioral: calorie health education knowledge and skills — 45 minute intervention done by health educator to give participants skills to use calorie information posted in fast-food restaurants
  Arms: Intervention

SUMMARY:
Increased consumption of fast-food may be a contributing factor to the obesity epidemic. Posting calories on menus in fast-food restaurants is an important public health initiative and may help consumers to make lower calorie, healthier choices. This study will develop and test an intervention to improve the impact of calorie labeling policies. Further, the study will examine potential barriers to using posted calorie information

DETAILED DESCRIPTION:
By the year 2030, 50% of American adults could be obese. Increasingly, Americans are consuming more foods away from home and most of these foods are consumed in fast-food restaurants. Menu calorie labeling provides calorie information at the point of purchase in fast-food restaurants and is one strategy employed to promote lower calorie, healthier food choices. Initial studies of the impact of calorie labeling, however, suggest that posting calories may only affect calories purchased in a minority of consumers.

The Patient Protection and Affordable Care Act (PPACA) mandates that calorie labeling be implemented nationally and fast-food restaurants throughout the U.S. will begin to post calorie information. With an overarching goal of improving the impact of calorie labeling policies; this proposal will develop and pilot test a brief intervention that is complementary to the posted calorie information, and will explore potential barriers to reducing calories among an urban clinic population. The study aims are: (Aim 1) To develop the Complementary Calorie Labeling (CCL) intervention, an individual single-session intervention that can be delivered in primary care settings. Semi-structured interviews will be conducted among 40 overweight or obese participants to guide development of intervention components and materials. (Aim 2) To conduct a pilot randomized controlled trial of the CCL intervention among 188 overweight or obese participants. The CCL intervention will be compared to a control group that receives an educational brochure about calories. The primary outcome will be weekly calories purchased at fast-food restaurants as measured by fast-food receipts and food logs. (Aim 3) To examine whether calorie knowledge, health literacy, numeracy, and motivation are barriers to using calorie information and whether these variables moderate intervention efficacy.

The proposed study will be conducted in a primarily low-income, minority clinic population in the Bronx NYC. NYC was the first major city to implement calorie labeling. Preliminary data from NYC suggest that fast-food consumers in the Bronx may be less likely to reduce their calories purchased when calorie information is posted, compared to other consumers in NYC. Developing interventions that may improve the impact of calorie labeling policies within this population will have important implications as these policies are implemented in urban communities throughout the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Eats at Fast-food restaurant at least once per week BMI>25

Exclusion Criteria:

* inability to keep food logs or fast-food receipts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
fast-food calories per week | 4 weeks
  change in fast-food calories purchased

CONTACTS AND LOCATIONS:
Overall Officials: Nichola Davis, Principal Investigator — New York City Health and Hospitals Corporation

IPD SHARING:
Plan to Share IPD: No